CLINICAL TRIAL: NCT00646932
Title: A Phase 2, Open-Label, Multicenter, Multi-Dose Study to Evaluate the Pharmacokinetics and Tolerability of Paricalcitol Injection in Chronic Kidney Disease Stage 5 Subjects With Secondary Hyperparathyroidism Undergoing Hemodialysis
Brief Title: Paricalcitol Injection Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Yoshihiko Ueki, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: J-ZEM-05-002
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: paricalcitol
- 2 (Experimental)
  Interventions: Drug: paricalcitol
- 3 (Experimental)
  Interventions: Drug: paricalcitol
- 4 (Experimental)
  Interventions: Drug: paricalcitol

INTERVENTIONS:
Drug: paricalcitol — paricalcitol 0.04 mcg/kg three times a week
  Other Names: ABT-358; Zemplar
  Arms: 1
Drug: paricalcitol — paricalcitol 0.08 mcg/kg three times a week
  Other Names: ABT-358; Zemplar
  Arms: 2
Drug: paricalcitol — paricalcitol 0.16 mcg/kg three times a week
  Other Names: ABT-358; Zemplar
  Arms: 3
Drug: paricalcitol — paricalcitol 0.24 mcg/kg three times a week
  Other Names: ABT-358; Zemplar
  Arms: 4

SUMMARY:
The PK and tolerability of paricalcitol after repeated intravenous administration for 2 weeks (total 6 doses at every HD session) are studied in subjects with 2°HPT who are receiving HD 3 times a week for stable chronic renal failure.

DETAILED DESCRIPTION:
The purpose of this study is pharmacokinetic & tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 2°HPT who are receiving HD 3 times a week for stable chronic renal failure

Exclusion Criteria:

* Subject is considered by investigator, for any reason, to be an unsuitable candidate for the study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 2 weeks

SECONDARY OUTCOMES:
Safety | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hideaki Harada, Study Director — Abbott
Locations (10):
- Japan (10):
  - Gunma
  - Hokkaido
  - Ibaraki
  - Kagoshima
  - Kumamoto
  - Nagano
  - Nagasaki
  - Saitama
  - Shizuoka
  - Tokyo